CLINICAL TRIAL: NCT01006603
Title: A 52-Week, Randomised, Double Blind, Active-Controlled, Multi-Centre Phase IIIb/IV Study to Evaluate the Efficacy and Tolerability of Saxagliptin Compared to Glimepiride in Elderly Patients With Type 2 Diabetes Mellitus Who Have Inadequate Glycaemic Control on Metformin Monotherapy
Brief Title: Saxagliptin Compared to Glimepiride in Elderly Type 2 Diabetes Patients, With Inadequate Glycemic Control on Metformin
Acronym: GENERATION
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D1680L00002
Record Dates: First submitted 2009-10-31; First posted 2009-11-03 (Estimated); Results first posted 2013-11-28 (Estimated); Last update posted 2013-11-28 (Estimated); Status verified 2013-09

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus; elderly patients; saxagliptin; randomised; double-blind
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — saxagliptin; glimepiride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Saxagliptin 5 mg
  Interventions: Drug: Saxagliptin
- 2 (Active Comparator): Glimepiride 1 - 6 mg
  Interventions: Drug: Glimepiride

INTERVENTIONS:
Drug: Saxagliptin — 5 mg, oral tablet, once daily
  Other Names: Onglyza
  Arms: 1
Drug: Glimepiride — 1, 2, 3, 4 or 6 mg, oral encapsulated tablet, once daily
  Other Names: Amaryl
  Arms: 2

SUMMARY:
This study will evaluate the efficacy and tolerability of saxagliptin compared to glimepiride in elderly patients with type 2 diabetes mellitus who have inadequate glycaemic control on metformin monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures
* Established clinical diagnosis of type 2 diabetes. Treatment with a stable metformin monotherapy, for at least 8 weeks prior to Visit 1
* HbA1c ≥7.0% and ≤9.0%

Exclusion Criteria:

* Type 1 diabetes, history of diabetic ketoacidosis or hyperosmolar non-ketonic coma. Current use of any injectable or oral antihyperglycemic agent excluding metformin.
* Renal impairment as defined by a creatinine clearance <60 mL/min
* Individuals who, in the opinion of the investigator, in which participation in this study may pose a significant risk to the patient and could render the patient unable to successfully complete the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 957 (Actual)
Dates: Start 2009-10; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (131):
- Austria (4):
  - Research Site, Feldbach
  - Research Site, Graz
  - Research Site, Salzburg
  - Research Site, Vienna
- Denmark (10):
  - Research Site, Aalborg
  - Research Site, Ans
  - Research Site, Kjellerup
  - Research Site, Kolding
  - Research Site, Nørresundby
  - Research Site, Roskilde
  - Research Site, Roslev
  - Research Site, Viborg
  - Research Site, Viby J
  - Research Site, Værløse
- Finland (12):
  - Research Site, Lahti, Finland
  - Research Site, Vantaa, Finland
  - Research Site, Harjavalta
  - Research Site, Helsinki
  - Research Site, Kuopio
  - Research Site, Kuusankoski
  - Research Site, Oulu
  - Research Site, Seinäjoki
  - Research Site, Sipoo
  - Research Site, Tampere
  - Research Site, Turku
  - Research Site, Vimpeli
- France (7):
  - Research Site, Châtellerault
  - Research Site, La Rochelle
  - Research Site, La Seyne-sur-Mer
  - Research Site, Laval
  - Research Site, Seysses
  - Research Site, Strasbourg
  - Research Site, Tiercé
- Germany (16):
  - Research Site, Hamburg, Hamburg
  - Research Site, Augsburg
  - Research Site, Darmstadt
  - Research Site, Dresden
  - Research Site, Essen
  - Research Site, Gelnhausen
  - Research Site, Hamburg
  - Research Site, Magdeburg
  - Research Site, Mayen
  - Research Site, München
  - Research Site, Neumünster
  - Research Site, Nuremberg
  - Research Site, Pirna
  - Research Site, Ratzeburg
  - Research Site, Reinfeld
  - Research Site, Sulzbach
- Greece (4):
  - Research Site, Athens, Greece
  - Research Site, Athens
  - Research Site, Nikaia
  - Research Site, Thessaloniki
- Hungary (6):
  - Research Site, Ács
  - Research Site, Balatonfüred
  - Research Site, Budapest
  - Research Site, Érd
  - Research Site, Gyöngyös
  - Research Site, Komárom
- Italy (9):
  - Research Site, Milan, MI
  - Research Site, Palermo, PA
  - Research Site, Padua, PD
  - Research Site, Pordenone, PN
  - Research Site, Reggio Emilia, RE
  - Research Site, Chieti
  - Research Site, Napoli
  - Research Site, Roma
  - Research Site, Viterbo
- Mexico (3):
  - Research Site, Durango, Durango
  - Research Site, Guadalajara, Jalisco
  - Research Site, Monterrey, Nuevo León
- Norway (18):
  - Research Site, Aksdal
  - Research Site, Ålesund
  - Research Site, Elverum
  - Research Site, Halden
  - Research Site, Hamar
  - Research Site, Kirkenær
  - Research Site, Kongsvinger
  - Research Site, Larvik
  - Research Site, Lierskogen
  - Research Site, Nordlenangen
  - Research Site, Oslo
  - Research Site, Røa
  - Research Site, Sandvika
  - Research Site, Skedsmokorset
  - Research Site, Svelvik
  - Research Site, Sørumsand
  - Research Site, Trondheim
  - Research Site, Ulset
- Spain (9):
  - Research Site, Seville, Andalusia
  - Research Site, Zamora, Castille and León
  - Research Site, A Coruña, Galicia
  - Research Site, Begonte (lugo), Galicia
  - Research Site, Getafe, Madrid
  - Research Site, Madrid, Madrid
  - Research Site, San Sebastián de los Reyes, Madrid
  - Research Site, Oviedo, Principality of Asturias
  - Research Site, Alicante, Valencia
- Sweden (13):
  - Research Site, Jönköping, Sweden
  - Research Site, Finspång
  - Research Site, Gävle
  - Research Site, Gothenburg
  - Research Site, Jarfalla
  - Research Site, Lessebo
  - Research Site, Lund
  - Research Site, Ödeshög
  - Research Site, Piteå
  - Research Site, Rättvik
  - Research Site, Stockholm
  - Research Site, Trollhättan
  - Research Site, Västervik
- United Kingdom (20):
  - Research Site, Fowey, Cornwall
  - Research Site, Nr Penzance, Cornwall
  - Research Site, Penzance, Cornwall
  - Research Site, Barnstaple, Devon
  - Research Site, Plymouth, Devon
  - Research Site, Annan, Dumfries and Galloway
  - Research Site, Canterbury, Kent
  - Research Site, Whitstable, Kent
  - Research Site, Frome, Somerset
  - Research Site, Bradford-on-Avon, Wiltshire
  - Research Site, Trowbridge, Wiltshire
  - Research Site, Ayrshire
  - Research Site, Bath
  - Research Site, Cumbernauld
  - Research Site, Dundee
  - Research Site, Hamilton
  - Research Site, Middlesex
  - Research Site, Motherwell
  - Research Site, Somerset
  - Research Site, Wellingborough

REFERENCES:
- [Derived] Perl S, Cook W, Wei C, Ohman P, Hirshberg B. Effects of Glimepiride versus Saxagliptin on beta-Cell Function and Hypoglycemia: A Post Hoc Analysis in Older Patients with Type 2 Diabetes Inadequately Controlled with Metformin. Clin Ther. 2016 Dec;38(12):2578-2588. doi: 10.1016/j.clinthera.2016.10.006. Epub 2016 Nov 4. PMID 27823868
- [Derived] Schernthaner G, Duran-Garcia S, Hanefeld M, Langslet G, Niskanen L, Ostgren CJ, Malvolti E, Hardy E. Efficacy and tolerability of saxagliptin compared with glimepiride in elderly patients with type 2 diabetes: a randomized, controlled study (GENERATION). Diabetes Obes Metab. 2015 Jul;17(7):630-8. doi: 10.1111/dom.12461. Epub 2015 Apr 7. PMID 25761977

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In total, 152 study centres in 13 countries recruited patients in this study. The first patient was enrolled in the study on 20 October 2009, and the last patient completed the study on 14 June 2012. 957 subjects were enrolled. 753 were deemed eligible for lead-in and 720 were randomized.
Pre-assignment Details: A 2-week single-blind (to patient only) placebo lead-in period occurred from Week -2 to Week 0. Patients were from this period on,counselled on dietary and lifestyle modifications according to usual clinical routine. They were given a glucometer to check their plasma glucose at home at least every second day.
Groups:
- Saxagliptin 5 mg: Saxagliptin 5 mg, oral tablet, once daily
- Glimepiride 1 - 6 mg: Glimepiride : 1, 2, 3, 4 or 6 mg, oral encapsulated tablet, once daily
Period: Overall Study
Arm/Group | Saxagliptin 5 mg | Glimepiride 1 - 6 mg
Started | 360 (Completed lead-in period and were randomised) | 360 (Completed lead-in period and were randomised)
Completed | 289 | 285
Not Completed | 71 | 75
Not completed — Withdrawal by Subject | 17 | 19
Not completed — Lost to Follow-up | 0 | 1
Not completed — Safety reason | 1 | 1
Not completed — Protocol Violation | 1 | 3
Not completed — Incorrect enrolment | 0 | 2
Not completed — Adverse Event | 15 | 7
Not completed — Death | 1 | 1
Not completed — Study specific discontinuation criteria | 33 | 34
Not completed — Other | 3 | 7

BASELINE CHARACTERISTICS:
Groups:
- Glimepiride 1 - 6 mg: Glimepiride 1, 2, 3, 4 or 6 mg, oral encapsulated tablet, once daily
- Total: Total of all reporting groups
Arm/Group | Saxagliptin 5 mg | Glimepiride 1 - 6 mg | Total
Number analyzed (Participants) | 360 | 360 | 720
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 360 | 360 | 720
Age Continuous [Mean (Standard Deviation); unit: years] | 72.5 (5.72) | 72.7 (5.44) | 72.6 (5.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 143 | 132 | 275
  Male | 217 | 228 | 445
Region of Enrollment [Number; unit: participants]
  Greece | 21 | 18 | 39
  Finland | 24 | 19 | 43
  Spain | 31 | 25 | 56
  Austria | 30 | 15 | 45
  United Kingdom | 39 | 49 | 88
  Italy | 12 | 12 | 24
  France | 11 | 13 | 24
  Hungary | 9 | 9 | 18
  Mexico | 10 | 7 | 17
  Denmark | 16 | 17 | 33
  Germany | 44 | 55 | 99
  Norway | 47 | 59 | 106
  Sweden | 66 | 62 | 128

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Reaching HbA1c <7% After 52 Weeks of Treatment Without Confirmed or Severe Hypoglycaemia.
Description: Defined as obtained on or before the 8th day after the last dosing day, as determined by central laboratory. Safety analysis set.
  Confirmed hypoglycaemia defined as: any event defined as either a symptomatic event with blood glucose level <3 mmol/L (<54 mg/dL) and no need for external assistance, or an asymptomatic blood glucose measurement <3 mmol/L (<54 mg/dL).
  Major (or severe) hypoglycaemia defined as: symptomatic events requiring external assistance due to severe impairment in consciousness or behaviour, with or without blood glucose level <3 mmol/L (<54 mg/dL), but with prompt recovery after glucose or glucagon administration. These events may be associated with sufficient neuroglycopenia to induce seizure or coma. Plasma glucose measurements may not be available during such an event, but neurological recovery, attributable to the restoration of plasma glucose to normal, was considered sufficient evidence that the event was induced by a low plasma glucose concentration.
Time Frame: From week 0 to week 52.
Population: Safety analysis set (a subset of the randomised analysis set including patients who took at least one investigational product dose).
Measure: Number; unit: percentage of participants
Arm/Group | Saxagliptin 5 mg | Glimepiride 1 - 6 mg
Number analyzed (Participants) | 359 | 359
percentage of participants
  All patients | 37.9 | 38.2
  patients aged <75 years (n=217, n=216) | 39.2 | 33.3
  patients aged ≥75 years (n=142, n=143) | 35.9 | 45.5

2. Secondary Outcome: Proportion of Patients Having Experienced at Least One Hypoglycaemic Event (Confirmed or Severe) Over the 52-week Double-blind Treatment Period.
Description: Hypoglyceamic event defined as, Confirmed hypoglycaemia: any event defined as either a symptomatic event with blood glucose level <3 mmol/L (<54 mg/dL) and no need for external assistance, or an asymptomatic blood glucose measurement <3 mmol/L (<54 mg/dL).
  Major (or severe) hypoglycaemia: symptomatic events requiring external assistance due to severe impairment in consciousness or behaviour, with or without blood glucose level <3 mmol/L (<54 mg/dL), but with prompt recovery after glucose or glucagon administration. These events may be associated with sufficient neuroglycopenia to induce seizure or coma. Plasma glucose measurements may not be available during such an event, but neurological recovery, attributable to the restoration of plasma glucose to normal, was considered sufficient evidence that the event was induced by a low plasma glucose concentration. Safety analysis set.
Time Frame: From week 0 to week 52.
Population: as for outcome 1
Measure: Number; unit: percentage of patients
Arm/Group | Saxagliptin 5 mg | Glimepiride 1 - 6 mg
Number analyzed (Participants) | 359 | 359
percentage of patients | 1.1 | 15.3

3. Secondary Outcome: Change From Baseline to Week 52 in HbA1c.
Description: Measured as the difference between the last on-treatment value (defined as obtained before or on the 8th day after the last dosing date), and the last pre-randomisation HbA1c value, as determined by central laboratory. Full analysis set.
Time Frame: From week 0 to week 52.
Population: The number of subjects with non-missing baseline and Week 52 (LOCF) values in the full analysis set (defined as the subset of patients in the randomized analysis set who took at least one randomised IP dose and have non-missing baseline and post-baseline efficacy data for at least one variable).
Measure: Mean (95% Confidence Interval); unit: % of glycosylated hemoglobin
Arm/Group | Saxagliptin 5 mg | Glimepiride 1 - 6 mg
Number analyzed (Participants) | 353 | 345
% of glycosylated hemoglobin | -0.44 [-0.51 to -0.37] | -0.64 [-0.71 to -0.57]

4. Secondary Outcome: Proportion of Patients Achieving a Therapeutic Glycaemic Response at Week 52 Defined as HbA1c <7.0%
Description: Proportion of patients with their last on-treatment value (defined as obtained before or on the 8th day after the last dosing date), as determined by central laboratory, below the specified limits. Full analysis set.
Time Frame: From week 0 to week 52
Population: as for outcome 3
Measure: Number; unit: percentage of responders
Arm/Group | Saxagliptin 5 mg | Glimepiride 1 - 6 mg
Number analyzed (Participants) | 356 | 353
percentage of responders | 44.7 | 54.7

5. Secondary Outcome: Change From Baseline to Week 52 in Fasting Plasma Glucose (FPG)
Description: Measured as the difference between the last on-treatment value (defined as obtained before or on the first day after the last dosing date)and the last pre-randomisation fasting plasma glucose value, as determined by central laboratory. Full analysis set.
Time Frame: From week 0 to week 52
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Saxagliptin 5 mg | Glimepiride 1 - 6 mg
Number analyzed (Participants) | 344 | 339
mmol/L | -0.73 [-0.89 to -0.57] | -1.29 [-1.45 to -1.13]

6. Secondary Outcome: Change From Baseline to Week 52 in Insulin
Description: Measured as the difference between the last on-treatment value (defined as obtained before or on the first day after the last dosing date) and the last pre-randomisation fasting plasma insulin value, as determined by central laboratory. Full analysis set.
Time Frame: From week 0 to week 52
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: µU/mL
Arm/Group | Saxagliptin 5 mg | Glimepiride 1 - 6 mg
Number analyzed (Participants) | 312 | 309
µU/mL | -2.0 [-3.1 to -1.0] | -0.6 [-1.6 to 0.5]

7. Secondary Outcome: Change From Baseline to Week 52 in β-cell Function (as Measured by Homeostasis Model Assessment-β [HOMA-β]
Description: β-cell function as estimated by the homeostasis model assessment (HOMA) model. Value is derived from FPG and fasting insulin; fasting insulin values below 2.074 μU/mL or above 57.595 μU/mL and FPG values below 3 mmol/L or above 25 mmol/L are excluded (as restricted by the calculation method used). Full analysis set.
Time Frame: From week 0 to week 52
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: percentage of change from baseline
Arm/Group | Saxagliptin 5 mg | Glimepiride 1 - 6 mg
Number analyzed (Participants) | 240 | 247
percentage of change from baseline | 3.83 [0.79 to 6.88] | 16.22 [13.23 to 19.20]

ADVERSE EVENTS:
Description: The at Risk population includes only those randomized subjects who took at least one dose of study drug.
Arm/Group | Saxagliptin 5 mg | Glimepiride 1 - 6 mg
Serious Adverse Events (participants affected / at risk) | 41/359 | 32/359
Other Adverse Events (participants affected / at risk) | 130/359 | 129/359
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Saxagliptin 5 mg (N=359) | Glimepiride 1 - 6 mg (N=359)
ANAEMIA (Blood and lymphatic system disorders) | 1 | 0
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 0 | 1
CARDIAC FAILURE (Cardiac disorders) | 1 | 3
MYOCARDIAL INFARCTION (Cardiac disorders) | 3 | 1
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 2
ATRIAL FIBRILLATION (Cardiac disorders) | 2 | 1
ANGINA PECTORIS (Cardiac disorders) | 1 | 1
ANGINA UNSTABLE (Cardiac disorders) | 1 | 0
ISCHAEMIC CARDIOMYOPATHY (Cardiac disorders) | 1 | 0
PERICARDITIS (Cardiac disorders) | 1 | 0
TACHYCARDIA (Cardiac disorders) | 0 | 1
EPIGASTRIC DISCOMFORT (Gastrointestinal disorders) | 1 | 0
HIATUS HERNIA (Gastrointestinal disorders) | 1 | 0
INGUINAL HERNIA (Gastrointestinal disorders) | 1 | 0
MELAENA (Gastrointestinal disorders) | 1 | 0
SUBILEUS (Gastrointestinal disorders) | 0 | 1
CHEST PAIN (General disorders) | 1 | 0
DEATH (General disorders) | 0 | 1
DEVICE DISLOCATION (General disorders) | 1 | 0
INFLAMMATION (General disorders) | 1 | 0
CHOLECYSTITIS (Hepatobiliary disorders) | 1 | 0
ANAPHYLACTIC SHOCK (Immune system disorders) | 1 | 0
PNEUMONIA (Infections and infestations) | 3 | 3
APPENDICITIS (Infections and infestations) | 1 | 0
DIVERTICULITIS (Infections and infestations) | 0 | 1
GASTROENTERITIS (Infections and infestations) | 0 | 1
GASTROENTERITIS NOROVIRUS (Infections and infestations) | 0 | 1
INFECTIOUS PLEURAL EFFUSION (Infections and infestations) | 0 | 1
LABYRINTHITIS (Infections and infestations) | 0 | 1
PYELONEPHRITIS (Infections and infestations) | 1 | 0
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1
URINARY TRACT INFECTION (Infections and infestations) | 0 | 1
UROSEPSIS (Infections and infestations) | 1 | 0
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 2 | 0
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
CONCUSSION (Injury, poisoning and procedural complications) | 1 | 0
CONTUSION (Injury, poisoning and procedural complications) | 0 | 1
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
HAND FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
MUSCLE RUPTURE (Injury, poisoning and procedural complications) | 0 | 1
MEDICAL OBSERVATION (Investigations) | 0 | 1
WEIGHT DECREASED (Investigations) | 1 | 0
HYPERKALAEMIA (Metabolism and nutrition disorders) | 1 | 0
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 | 1
JOINT EFFUSION (Musculoskeletal and connective tissue disorders) | 0 | 1
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
SPINAL COLUMN STENOSIS (Musculoskeletal and connective tissue disorders) | 1 | 0
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
BLADDER TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
BREAST CANCER IN SITU (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
HEPATIC NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
LUNG CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
PANCREATIC CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
SALIVARY GLAND CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 | 1
EPILEPSY (Nervous system disorders) | 0 | 1
SYNCOPE (Nervous system disorders) | 1 | 1
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 | 1
CALCULUS BLADDER (Renal and urinary disorders) | 1 | 0
CALCULUS URETERIC (Renal and urinary disorders) | 0 | 1
NEUROGENIC BLADDER (Renal and urinary disorders) | 0 | 1
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
SURGICAL AND MEDICAL PROCEDURES CARDIOVERSION Systematic Assessment 0 359 1 359 (Surgical and medical procedures) | 1 | 0
AORTIC ANEURYSM (Vascular disorders) | 1 | 0
AORTIC ARTERIOSCLEROSIS (Vascular disorders) | 0 | 1
CIRCULATORY COLLAPSE (Vascular disorders) | 0 | 1
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Saxagliptin 5 mg (N=359) | Glimepiride 1 - 6 mg (N=359)
VERTIGO (Ear and labyrinth disorders) | 9 | 0
DIARRHOEA (Gastrointestinal disorders) | 15 | 19
CONSTIPATION (Gastrointestinal disorders) | 4 | 10
NAUSEA (Gastrointestinal disorders) | 4 | 8
NASOPHARYNGITIS (Infections and infestations) | 23 | 35
URINARY TRACT INFECTION (Infections and infestations) | 11 | 18
BRONCHITIS (Infections and infestations) | 14 | 7
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 12 | 14
CONTUSION (Injury, poisoning and procedural complications) | 8 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 9 | 18
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 17 | 9
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 10 | 9
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 9 | 3
DIZZINESS (Nervous system disorders) | 6 | 17
HEADACHE (Nervous system disorders) | 6 | 12
TREMOR (Nervous system disorders) | 1 | 8
COUGH (Respiratory, thoracic and mediastinal disorders) | 9 | 13
HYPERTENSION (Vascular disorders) | 8 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication or presentation may include any of AZ's confidential information without AZ's prior written approval.